CLINICAL TRIAL: NCT01391091
Title: Effect of Catheter Ablation on the Prevalence, Clinical Manifestation and MRI Findings of Migraine in AF Patients With or Without a Previous History of Migraine
Brief Title: Effect of Catheter Ablation on Clinical Course of Migraine in AF Patients With or Without Previous History of Migraine
Acronym: CONFIRM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Texas Cardiac Arrhythmia Research Foundation (Other)
Responsible Party: Principal Investigator, Andrea Natale, Medical director, Texas Cardiac Arrhythmia Research Foundation
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TCAI-CONFIRM
Record Dates: First submitted 2011-05-26; First posted 2011-07-11 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2015-05

CONDITIONS: Migraine; Atrial Fibrillation
MeSH Terms: conditions — Migraine Disorders; Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients without history of migraine (Active Comparator): Incidence and prevalence of migraine episodes in the post-ablation period
  Interventions: Procedure: Radiofrequency catheter ablation
- Patients with history of migraine (Active Comparator): Incidence and prevalence of migraine episodes in the post-ablation period
  Interventions: Procedure: Radiofrequency catheter ablation

INTERVENTIONS:
Procedure: Radiofrequency catheter ablation — PVAI
  Other Names: AF ablation; Pulmonary Vein Antral Ablation
  Arms: Patients without history of migraine
Procedure: Radiofrequency catheter ablation — PVAI
  Other Names: AF ablation; Pulmonary Vein Antral Ablation
  Arms: Patients with history of migraine

SUMMARY:
The purpose of this prospective study is to evaluate the effect of catheter ablation on incidence, prevalence and disease-severity of migraine in AF patients undergoing ablation, with or without a history of migraine.

DETAILED DESCRIPTION:
Migraine, a neurovascular disorder affecting approximately 12% of world population, is characterized by recurrent attacks of incapacitating headache associated with photophobia, phonophobia, nausea and vomiting (1). Although the pathogenesis of migraine is not clearly understood yet, it has been widely accepted as being caused by cerebral vasodilatation, abnormal neurological firings and/or neurogenic dural inflammation (1). Additionally, recent studies have demonstrated an association between migraine with aura and intracardiac shunting by a patent foramen ovale (PFO) leading to a hypothesis that paradoxical brain embolism of platelets and other undefined chemical substances can play a causal role in migraine with aura (2).

Radiofrequency catheter ablation (RFCA) has been shown to be a promising treatment for cardiac arrhythmias. During catheter ablation, trans-septal puncture (TSP) is routinely performed to gain access to the left heart. TSP causes an iatrogenic atrial septal defect (ASD) with a transient right-to-left shunt which can predispose patients to stroke and migraine (3). In two different studies, with 571 and 183 patients in whom TSP was performed, the incidence of migraine was 0.5% and 2.2% respectively and the migraine was transient and resolved without any sequelae (2, 3). In separate studies, complete resolution or improvement of migraine was noticed with the ASD/PFO closure (4). Additional case-studies have also reported AF occurring during episodes of migraine with aura where the cardiac rhythm was normal between the episodes (5). All these reports evidently demonstrate an association between AF, TSP during RFCA and migraine, but fail to clearly define the nature of it. It is not yet understood whether a successful catheter ablation of AF has any impact on the natural course of pre-existing or newly-occurring migraine. This study aims at exploring the relationship between AF and migraine and to evaluate if an effective ablation therapy for AF influences the incidence and clinical presentation of migraine in patients with or without a previous history.

Several isolated case-studies have reported improvement in the frequency and severity of migraine during treatment with Coumadin (6, 7). Coumadin is routinely prescribed to patients undergoing RFCA to prevent thrombo-embolic events. Our study would further explore the impact of therapeutic Coumadin on the prevalence and clinical course of migraine in patients with a previous history.

Hypothesis: Catheter ablation affects the disease course of migraine in AF patients with or without a previous history of migraine.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-75 years
* AF patients undergoing RFCA
* Ability to distinguish migraine attacks as discrete from other headaches (i.e., tension-headache)
* Ability to read, comprehend, and legibly and reliably record information
* Ability to provide written, informed consent

Exclusion Criteria:

* Uncontrollable hypertension
* History of stroke, TIA or epilepsy
* Bleeding disorder
* Hypersensitivity, allergy or contraindications to the use of NSAIDs, Triptans, Aspirin or Warfarin
* Contraindication to undergoing an MRI

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2010-12; Primary Completion 2013-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Incidence of thrombo-embolic events and migraine | 6 and 12 months post-ablation

SECONDARY OUTCOMES:
Impact of therapeutic Coumadin on the prevalence and clinical course of migraine in patients with a previous history | 6 and 12 months post-ablation

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Natale, MD, Principal Investigator — Texas Cardiac Arrhythmia Research Foundation; Luigi Di Biase, MD, Phd, Principal Investigator — Texas Cardiac Arrhythmia Research Foundation
Locations (1):
- St. David's Medical Center, Austin, Texas, United States